CLINICAL TRIAL: NCT01221272
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Cross-over Trial to Evaluate the Effects of Ranolazine on Myocardial Perfusion Assessed by Serial Quantitative Exercise SPECT Imaging
Brief Title: Effect of Ranolazine on Myocardial Perfusion Assessed by Serial Quantitative Exercise SPECT Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-259-0103
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Myocardial Perfusion Imaging; Myocardial Ischemia
Keywords: SPECT MPI
MeSH Terms: conditions — Myocardial Ischemia | interventions — Ranolazine; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine/Placebo (Experimental): Participants received ranolazine from Day 1 through Day 15 (± 2 days) of Period 1, followed by an exercise SPECT MPI study, then received placebo to match ranolazine from Day 1 through Day 15 (± 2 days) of Period 2, followed by an exercise SPECT MPI study.
  Interventions: Drug: Ranolazine; Drug: Placebo to match ranolazine; Procedure: SPECT MPI; Behavioral: Exercise
- Placebo/Ranolazine (Experimental): Participants received placebo to match ranolazine from Day 1 through Day 15 (± 2 days) of Period 1, followed by an exercise SPECT MPI study, then received ranolazine from Day 1 through Day 15 (± 2 days) of Period 2, followed by an exercise SPECT MPI study.
  Interventions: Drug: Ranolazine; Drug: Placebo to match ranolazine; Procedure: SPECT MPI; Behavioral: Exercise

INTERVENTIONS:
Drug: Ranolazine — * One 500 mg tablet in the evening on Day 1 of the period
  * One 500 mg tablet, twice daily on Days 2-3 of the period
  * Two 500 mg tablets (1000 mg total), twice daily from Day 4 to the end of the period (Day 15 ± 2 days)
  Other Names: Ranexa®
Drug: Placebo to match ranolazine — Placebo to match ranolazine administered in the same form and frequency as the active drug.
Procedure: SPECT MPI — Gated single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) to confirm the presence of reversible exercise-induced left ventricular perfusion defect size (PDS) performed within 12 weeks prior to baseline or at the baseline visit, and at the end-of-period 1 and end-of-period 2 visits.
Behavioral: Exercise — Treadmill stress test

SUMMARY:
This study enrolled participants with documented exercise-induced myocardial ischemia in order to evaluate whether ranolazine, when taken prior to exercise, can improve blood flow to the heart (myocardial perfusion), as assessed by exercise-induced myocardial perfusion defect size (PDS) and total perfusion deficit (TPD), using gated single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI).

This was a 2-period crossover study. The last dose of each period must have been taken 3-4 hours prior to conduct of the exercise SPECT MPI. After the research exercise SPECT MPI was performed at the end of Period 1, participants discontinued the treatment they were randomized to for that period and began the other treatment in Period 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Exercise SPECT MPI study (stress and rest) showing at least 10% reversible myocardial ischemia (as confirmed by the core nuclear laboratory using Corridor4DM imaging software) performed not more than 12 weeks prior to screening, OR
* Exercise SPECT MPI study (stress and rest) conducted during screening (after consultation with the Medical Monitor and after informed consent was obtained) showing at least 10% reversible myocardial ischemia (as confirmed by the core nuclear laboratory)
* Stable antianginal medical therapy (excluding short-acting nitroglycerin)

Key Exclusion Criteria:

* Left bundle branch block
* Automated implantable defibrillator and/or pacemaker (selected subjects with permanent pacemakers who had an intact sinus mechanism may have been included following consultation with the Medical Monitor)
* Intervening coronary revascularization between the time of qualifying exercise SPECT MPI study and randomization
* Acute myocardial infarction (MI) within 60 days prior to screening or at any time after the qualifying exercise SPECT MPI study, or MI undergoing staged intervention during a subject's participation in the trial
* Unstable angina within 30 days prior to screening, or at any time after the qualifying exercise SPECT MPI study
* Coronary artery bypass graft surgery within 60 days prior to screening or at any time after the qualifying exercise SPECT MPI study, or percutaneous coronary intervention within 30 days prior to screening or at any time after the qualifying exercise SPECT MPI study
* Anticipated coronary revascularization during the trial period
* Cerebrovascular attack or transient ischemic attack within 90 days prior to screening
* History of serious arrhythmias
* Current atrial fibrillation or atrial flutter
* QTc interval > 500 milliseconds
* Diagnosed as having New York Heart Association Class III or IV heart failure
* Inability to exercise or exercise limitation due to other comorbidities that may have interfered with ability to perform required exercise SPECT MPI study
* Body mass index greater than or equal to 38 kg/m^2 (may have been up to 40 kg/m^2 after consultation with the Medical Monitor)
* Any absolute contraindications to exercise stress testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yue, MD, Study Director — Gilead Sciences
Locations (43):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Imperial Cardiac Center, Imperial, California
  - Clinical Trials Research, Lincoln, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Central Coast Cardiology, Salinas, California
  - Alfieri Cardiology, Newark, Delaware
  - St. Luke's Cardiology Associates, Jacksonville, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Research One, Orlando, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Research Integrity, LLC, Owensboro, Kentucky
  - Louisiana Heart Center, Covington, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Androscroggin Cardiology Associates DBA Maine Research Associates, Auburn, Maine
  - Delmarva Heart Research Foundation, Inc, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cardiovascular Imaging Technologies, Kansas City, Missouri
  - Dr. Michael Sacher, Massapequa, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Heritage Cardiology, Camp Hill, Pennsylvania
  - University of Pittsburgh Medical Center Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Kore Cardiovascular Research, Jackson, Tennessee
  - East Texas Cardiology PA, Houston, Texas
  - Mercury Medical, LLC, San Antonio, Texas
- Canada (4):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - ECOGENE-21 Clinical Trial Center, Chicoutimi Hospital, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Chum Hotel Dieu, Montreal, Quebec
- Czechia (2):
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- Turku University Hospital, Turku, Finland
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Kaplan Medical Center, Rehovot
  - Assuta MC, Tel Aviv
- Italy (2):
  - "Federico II" University, Naples
  - Federico II University, Naples
- Singapore (2):
  - National University Health System, Singapore
  - National Heart Centre Singapore, Singapore
- Northwick Park Hospital, Watford Road, Middlesex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 27 study sites in the United States, Canada, Czech Republic, and Israel. The first participant was screened on 29 September 2010. The last participant observation was on 27 September 2012.
Pre-assignment Details: Number screened: 222; randomized and treated (RAT; Safety Analysis Set): 81
  Efficacy Analysis Set: 61 RAT participants with data for both end-of-period (EOP) scans, completed ≥ 7 consecutive days treatment in each period, took the morning dose before each EOP scan, and had baseline perfusion defect size ≥ 5% as measured by QPS imaging software.
Groups:
- Ranolazine/Placebo: Period 1: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise gated single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) study.
  Period 2: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
- Placebo/Ranolazine: Period 1: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Period 2: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
Period: Period 1
Arm/Group | Ranolazine/Placebo | Placebo/Ranolazine
Started | 41 | 40
Completed | 39 | 38
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Consent Withdrawal | 0 | 1
Not completed — Significant Dosing Noncompliance | 0 | 1
Period: Period 2
Arm/Group | Ranolazine/Placebo | Placebo/Ranolazine
Started | 39 | 39 (1 participant did not complete Period 1, but started and completed Period 2.)
Completed | 39 | 37
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- All Participants: Baseline characteristics were analyzed as a single group (Safety Analysis Set). All participants were assigned to complete the same treatment periods in the same manner.
  Ranolazine Treatment Period: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Placebo Treatment Period: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
Arm/Group | All Participants
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.0)
Age, Customized [Number; unit: participants]
  18 to 39 years | 0
  40 to 64 years | 29
  65 to 74 years | 39
  ≥ 75 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 75
Race/Ethnicity, Customized [Number; unit: participants]
  White | 72
  African-American | 5
  Other | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic Or Latino | 9
  Not Hispanic Or Latino | 62
  Not Reported | 5
  Unknown | 5
Region of Enrollment [Number; unit: participants]
  United States | 38
  Czech Republic | 2
  Canada | 27
  Israel | 14
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (3.8)
Weight [Mean (Standard Deviation); unit: kg] | 88.6 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Exercise-induced Perfusion Defect Size (PDS) Following Ranolazine and Placebo Treatment
Description: PDS is the amount (percent) of the myocardium with decreased blood flow. A lower percentage means more of the myocardium is receiving blood flow. Measurements were obtained by gated single photon emission computed tomography (SPECT) imaging following exercise at the end of the ranolazine and placebo treatment periods.
Time Frame: Up to 33 days
Population: Efficacy Analysis Set: 61 randomized and treated participants with data for both end-of-period (EOP) scans, completed ≥ 7 consecutive days treatment in each period, took the morning dose before each EOP scan, and had baseline perfusion defect size ≥ 5% as measured by QPS imaging software
Measure: Least Squares Mean (Standard Error); unit: percentage of myocardium
Groups:
- Ranolazine: Ranolazine treatment period: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
- Placebo: Placebo treatment period: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 61 | 61
percentage of myocardium | 21.54 (1.51) | 20.87 (1.51)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — The null hypothesis that ranolazine treatment had no effect on PDS would be rejected if the PDS and TPD p-values were less than 0.05 or the PDS p-value was less than 0.05/2 = 0.025; Mixed Models Analysis = 0.67, 95% CI 2-sided [-0.6 to 1.9]

2. Primary Outcome: Exercise-induced Total Perfusion Deficit (TPD) Following Ranolazine and Placebo Treatment
Description: TPD is a score that measures the overall impact of a region of decreased myocardial blood flow, incorporating both the amount and severity of the decreased flow. TPD is measured on a scale of 0-100, with higher scores being worse and lower scores being better. Measurements were obtained by SPECT imaging following exercise at the end of the ranolazine and placebo treatment periods.
Time Frame: Up to 33 days
Population: Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 61 | 61
units on a scale | 17.23 (1.26) | 16.57 (1.26)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.22, Mixed Models Analysis — The null hypothesis that ranolazine treatment had no effect on TPD would be rejected if the PDS and TPD p-values were less than 0.05 or the TPD p-value was less than 0.05/2 = 0.025; Mixed Models Analysis = 0.65, 95% CI 2-sided [-0.4 to 1.7]

3. Secondary Outcome: Perfusion Defect Severity at Baseline, End of Period 1, and End of Period 2
Description: Perfusion defect severity was assessed for each participant as the percentage of the 17 myocardium segments with a relative perfusion defect score of 3 or 4 on a 0-4 scale. Segment scores are: 0 = normal perfusion; 1 = mild reduction in counts-not definitely abnormal; 2 = moderate reduction in counts-definitely abnormal; 3 = severe reduction in counts; 4 = absent uptake (lower scores correspond to less severity and higher scores correspond to increased severity). A lower percentage means fewer segments have severely reduced blood flow. Measurements were obtained by SPECT imaging following exercise at baseline and at the end of Periods 1 and 2.
Time Frame: Up to 33 days
Population: Efficacy Analysis Set
Measure: Mean (Standard Error); unit: percentage of segments
Groups:
- Ranolazine/Placebo: Period 1: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Period 2: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
Arm/Group | Ranolazine/Placebo | Placebo/Ranolazine
Number analyzed (Participants) | 30 | 31
percentage of segments
  Baseline | 11.4 (2.0) | 8.5 (2.0)
  End of Period 1 | 11.6 (1.9) | 10.2 (2.1)
  End of Period 2 | 10.4 (1.9) | 9.5 (2.0)

4. Secondary Outcome: Exercise-induced Reversible Perfusion Defect Size (PDS) at Baseline, End of Period 1, and End of Period 2
Description: Exercise-induced reversible PDS was derived as the exercise PDS at baseline and at the end of Periods 1 and 2 minus the resting PDS at baseline. A lower percentage means more of the myocardium is receiving blood flow. Measurements were obtained by SPECT imaging at baseline both at rest and following exercise and following exercise at the end of Periods 1 and 2.
Time Frame: Up to 33 days
Population: Efficacy Analysis Set
Measure: Mean (Standard Error); unit: percentage of myocardium
Arm/Group | Ranolazine/Placebo | Placebo/Ranolazine
Number analyzed (Participants) | 30 | 31
percentage of myocardium
  Baseline exercise minus baseline resting | 12.5 (1.1) | 13.5 (1.3)
  End of Period 1 exercise minus baseline resting | 12.7 (1.2) | 14.1 (1.4)
  End of Period 2 exercise minus baseline resting | 12.4 (1.0) | 15.2 (1.4)

5. Secondary Outcome: Exercise-induced Reversible Total Perfusion Deficit (TPD) at Baseline, End of Period 1, and End of Period 2
Description: Exercise-induced reversible TPD was derived as the exercise TPD at baseline and at the end of Periods 1 and 2 minus the resting TPD at baseline. TPD is measured on a scale of 0-100, with higher scores being worse and lower scores being better. Measurements were obtained by SPECT imaging at baseline both at rest and following exercise and following exercise at the end of Periods 1 and 2.
Time Frame: Up to 33 days
Population: Efficacy Analysis Set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ranolazine/Placebo | Placebo/Ranolazine
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline exercise minus baseline resting | 10.5 (0.9) | 10.5 (1.0)
  End of Period 1 exercise minus baseline resting | 10.5 (0.9) | 10.7 (1.0)
  End of Period 2 exercise minus baseline resting | 10.1 (0.8) | 11.6 (1.1)

ADVERSE EVENTS:
Time Frame: Up to 33 days
Description: All participants were assigned to complete the ranolazine and placebo treatment periods during the study, the only difference being which treatment period they started first.
Groups:
- Onset Following Ranolazine: This reporting group includes participants dosed with ranolazine and their events for which the last dosed treatment was ranolazine, ie, events with onset during the ranolazine treatment period or during post-ranolazine treatment period follow-up.
  Ranolazine Treatment Period: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Placebo Treatment Period: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
- Onset Following Placebo: This reporting group includes participants dosed with placebo and their events for which the last dosed treatment was placebo, ie, events with onset during the placebo treatment period or during post-placebo treatment period follow-up.
  Ranolazine Treatment Period: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Placebo Treatment Period: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
- Onset at Any Time Following Ranolazine: This reporting group includes participants dosed with ranolazine and their events with onset at any time following ranolazine treatment.
  Ranolazine Treatment Period: Participants received ranolazine 1 × 500 mg tablet administered once in the evening on Day 1, 1 × 500 mg tablet twice daily on Days 2-3, and 2 × 500 tablets twice daily from Day 4 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
  Placebo Treatment Period: Participants received placebo to match ranolazine from Day 1 to the end of the period (Day 15 ± 2 days), followed by an exercise SPECT MPI study.
Arm/Group | Onset Following Ranolazine | Onset Following Placebo | Onset at Any Time Following Ranolazine
Serious Adverse Events (participants affected / at risk) | 2/80 | 0/79 | 2/80
Other Adverse Events (participants affected / at risk) | 25/80 | 7/79 | 28/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Onset Following Ranolazine (N=80) | Onset Following Placebo (N=79) | Onset at Any Time Following Ranolazine (N=80)
Bronchitis (Infections and infestations) | 1 | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Onset Following Ranolazine (N=80) | Onset Following Placebo (N=79) | Onset at Any Time Following Ranolazine (N=80)
Angina pectoris (Cardiac disorders) | 3 | 1 | 4
Constipation (Gastrointestinal disorders) | 6 | 1 | 6
Nausea (Gastrointestinal disorders) | 5 | 2 | 5
Dizziness (Nervous system disorders) | 11 | 0 | 11
Headache (Nervous system disorders) | 3 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years